CLINICAL TRIAL: NCT05222035
Title: Camrelizumab Plus PEG-rhG-CSF in Recurrent/Metastatic NPC With First-line Treatment Failure
Brief Title: PD-1 Inhibitor Plus G-CSF in Recurrent/Metastatic NPC With First-line Treatment Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Chief physician, Proffessor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-2021-1215
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: PD-1 Inhibitor; G-CSF
MeSH Terms: interventions — camrelizumab; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-CSF+Camrelizumab (Experimental)
  Interventions: Drug: Camrelizumab; Drug: G-CSF
- Camrelizumab (Active Comparator)
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — PD-1 inhibitor: Camrelizumab, 200 mg, intravenously (IV) , Day 1, Q3W, until progressive disease (PD) or unacceptable toxicity for a maximum of up to 35 cycles (up to approximately 2 years).
Drug: G-CSF — G-CSF: mecapegfilgrastim, 6 mg, subcutaneous injection, Day 1, Q3W, until stop using Camrelizumab, progressive disease (PD) or unacceptable toxicity.
  Arms: G-CSF+Camrelizumab

SUMMARY:
Recurrence and metastasis are the main causes of treatment failure of NPC. Preliminary clinical studies have found that the overall response rate of PD-1 inhibitors in treating ≥2 line R/M NPC is about 25%.

Recent studies have shown that G-CSF can significantly increase the proportion of effector cells dominated by CD4+ T cells, improve the diversity of peripheral blood TCR, and regulate the immune status of patients. Therefore, we suspect that G-CSF may have a synergistic effect on PD-1 inhibitor, thus enhance the efficacy of PD-1 inhibitor monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; 18-75 years of age.
2. Received one or more lines of therapy, which must include prior treatment with a platinum agent (except for patients who are unfit or refuse platinum-containing regimens) and must not be amenable to potentially curative radiotherapy or surgery. [Received neoadjuvant/adjuvant/concurrent platinum-containing regimen for radical therapy (radiotherapy or surgery), with recurrence ≤6 months following completion of therapy can be recognized as one line]
3. Subjects diagnosed with pathological confirmed non-keratinizing (WHO-II/III) metastatic NPC, or subjects with recurrent NPC that is unfit for local treatment
4. Patients must have at least 1 lesion that is measurable using RECIST v1.1 criteria.
5. ECOG performance status of 0 or 1.
6. Have recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to any anti-tumor therapy 4 weeks earlier. Except for hair loss, hair color change, nail change, fatigue, etc., which do not pose safety risks to subjects.
7. Life expectancy more than 12 weeks.
8. Patients must have adequate organ function (without blood transfusion, without growth factor or blood components support within 14 days before enrollment) as determined by:

   Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet count ≥ 75×109/L; Hemoglobin ≥ 9 g/dL; serum total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×upper limit of normal (ULN), (for subjects with liver metastases, TBIL ≤3×ULN ; ALT and AST≤5×ULN); Creatinine ≤1.5×ULN or creatinine clearance rate≥50 ml/min (Cockcroft-Gault formula); serum albumin ≥28 g/L; INR, APTT≤1.5 x ULN.
9. Female subjects agree not to be pregnant or lactating from beginning of the study screening through at least 3 months after receiving the last dose of study treatment. Both men and women of reproductive potential must be willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy.
10. Be willing and able to provide written informed consent/assent for the trial.

Exclusion Criteria:

1. Subjects who underwent anti-PD-1 /PD-L antibody or anti-CTLA-4 antibody (or any other antibody acting on T cell synergistic stimulation or checkpoint pathway).
2. Known history of hypersensitivity to any components of the Camrelizumab and PEG-rhG -CSF formulation or other monoclonal antibodies.
3. Prior chemotherapy, targeted small molecule therapy, or radical therapy within 2 weeks prior to Study Day 1
4. Diagnosed and/or treated additional malignancy within 5 years of enrollment, with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin, and/or curatively-resected in situ cervical and/or breast carcinoma.
5. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration.
6. Active central nervous system metastases and/or carcinomatous meningitis
7. Severe, uncontrolled angiocardiopathy (heart failure > class II NYHA, unstable angina, myocardial infarction within past 1 year, supraventricular or ventricular arrhythmia which need medical intervention, or QT interval male ≥ 450 ms, female ≥ 470 ms.).
8. History of non-infectious pneumonitis that required steroids or current pneumonitis
9. Active infection requiring systemic therapy
10. Be known to have active tuberculosis.
11. Human immunodeficiency virus (HIV) positive
12. Hepatitis B or C positive
13. Live vaccine within 30 days of planned start of study drug
14. Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-01-24 (Estimated); Primary Completion 2022-12-24 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 1 year
  Defined as the proportion of patients whose tumors shrink to complete response (CR) or partial response (PR) and remain for a certain period of time according to RECIST 1.1

SECONDARY OUTCOMES:
The proportion of patients who achieved disease control | 1 year
  Defined as the proportion of subjects who achieve CR+PR+stable disease (SD) for at least 4 weeks according to RECIST 1.1.
The proportion of patients who achieved clinical benefit | 1 year
  Defined as maintaining the efficacy of CR+PR+SD for at least 6 months according to RECIST 1.1.
median progression-free survival | 1 year
  Defined as the period from the start of enrollment until disease progression or death from any cause.
Duration of response | 1 year
  Defined as the time from the first assessment of CR and PR to the first assessment of PD or death caused by any cause according to RECIST 1.1.
Adverse events | 1 year
  assessed by NCI-CTC5.0 standard

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China